CLINICAL TRIAL: NCT01486472
Title: Lacrimal Drainage Obstruction in Gastric Cancer Patients Receiving Adjuvant S-1 Chemotherapy: A Prospective Study
Brief Title: S-1-induced Lacrimal Drainage Obstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Keun-Wook Lee, Clinical professor, Seoul National University Bundang Hospital
Other Study IDs: GC-SNUBH-2010-01; GC-CTX-01 (Other: SNUBH)
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Gastric Cancer
Keywords: Adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Tears
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GC patients receiving adjuvant S-1 chemotherapy
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — Adjuvant S-1 chemotherapy will be performed to GC patients receiving curative D2 gastric surgery

SUMMARY:
S-1 is an effective drug in gastric cancer (GC) for palliative chemotherapy in Eastern and Western patients. Recently, S-1 has been also reported to be an effective adjuvant therapy for GC patients who received D2 surgery in Eastern Asian patients.

Recently, the development of lacrimal drainage obstruction (LDO) caused by S-1 has been reported from some case and small-sized studies. The incidence of developing LDO has been estimated to about 15~20% of patients receiving S-1 therapy in some retrospective studies. However, there is no prospective report on the incidence of LDO in patients receiving S-1 chemotherapy. Moreover, the mechanism of developing S-1-induced LDO has not been systemically studied until now. Suggested mechanism of LDO involves direct secretion of S-1 into the tear.

Therefore, this study was initiated to prospectively investigate the incidence of LDO in GC patients receiving adjuvant S-1 chemotherapy. In addition, the correlation between the development of LDO and the concentration of S-1 (or its metabolites) in tear and plasma will be explored. These results will help clinicians identify patients who are at high risk of developing S-1-associated LDO.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received curative (R0) surgery for GC
* Patients receiving adjuvant S-1 chemotherapy
* Patients with adequate major organ functions for chemotherapy
* Patient who have taken S-1 at least 7 days (for blood and tear sampling)

Exclusion Criteria:

* Patients who are not candidate for adjuvant S-1 chemotherapy
* Patients with previous history of LDO
* Patients with other opthalmologic disease who are not appropriate to be included in this study (i.e., patients using eyedrop medication; patients with dry eye whose tears cannot be sampled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving S-1 as an adjuvant chemotherapy after radial surgery (D2 dissection) for GC
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of LDO | The incidence of LDO (1 year)
  The cumulative incidence of LDO during the 1 year after adjuvant S1 chemotherapy will be analyzed

SECONDARY OUTCOMES:
Correlation between the concentration of S-1-related chemical compounds and the developement of LDO
  Correlation between the concentration of S-1-related chemical compounds (5-FU or other components) and the risk of developing LDO will be investigated. Plasma and tear samples will be aquired during the chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Wook Lee, M.D. & Ph.D., Principal Investigator — Department of Internal Medicine, Seoul National University Bundang Hospital; Namju Kim, M.D., Principal Investigator — Department of Opthalmology, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea